CLINICAL TRIAL: NCT04791670
Title: USABILITY OF AN INTERACTIVE HEALTH TECHNOLOGY FOR KIDNEY LIVING DONORS ASSESSMENT: TOWARDS A STANDARDIZED INFORMED PROCESS
Brief Title: eHealth Usability in Living Kidney Donation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Oulu (Other)
Responsible Party: Principal Investigator, Fernanda Ortiz, Nephrologist, Helsinki University Central Hospital
Other Study IDs: eHealth/HUS/501
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Living Kidney Donation
Keywords: eHealth; value-based healthcare
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey study — The surveys will include general data, the type of electronic devices in possession and the purpose of use. eHealth literacy will be assessed with the eHeals questionnaire. Platform's ease of use will be assessed with the System Usability Scale, and participants´ opinion about the digital path utility with six questions. These items will be answered with a Likert-scale. Finally, we added an open question for qualitative analysis.

SUMMARY:
Several web portals for patients are available, but an assessment of their performance is scarce. This is of particular interest among candidates for kidney living donation. A crucial aspect of living donation is to provide standardized information about the risks of the procedure. In 2019 it was launched a personalized digital care path for kidney living candidates, which contains information about the donation process and facilitates the communication between clinicians, transplant coordinators, and patients, enabling telemedicine.

We aim to investigate living donor candidates' experience with the Health Village web portal and the digital care path for living donor candidates. The secondary aim is to investigate their attitude of living donor candidates to eHealth services.

DETAILED DESCRIPTION:
Background. Several web portals for kidney patients are available, but an assessment of their performance is scarce. This is of particular interest among candidates for kidney living donation. A crucial aspect of living donation is to provide standardized information about the risks of the procedure. In Finland, the web portal Health Village contains general information about kidney diseases. In 2019 it was launched a personalized digital care path for kidney living candidates, which contains information about the donation process and facilitates the communication between clinicians, transplant coordinators, and patients, enabling telemedicine. The performance of this eHealth service has not yet been studied.

Objectives. to investigate living donor candidates' experience with the web portal Health Village and the digital care path for living donor candidates. The secondary aim is to investigate their attitude of living donor candidates to eHealth services.

Methods. A prospective cross sectional survey study. Participants will be all kidney donor candidates who have used the digital care path since its implementation in January 2019 up to 1.3.2021 (N=122). The surveys will include general data, the type of electronic devices in possession and the purpose of use. eHealth literacy will be assessed with the eHeals questionnaire. Platform's ease of use will be assessed with the System Usability Scale, and participants´ opinion about the digital path utility with six questions. These items will be answered with a Likert-scale. Finally, we added an open question for qualitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Living donor candidates from Helsinki area, from 2019 onwards

Exclusion Criteria:

* Living donor candidates from other areas of the country
* non-Finnish speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All living donor candidates who contacted the living donor transplant coordinator, and were considered initially suitable for kidney donation.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Patient´s experience | 4 months
  Measured with Likert scale
Patient´s e-Health literature | 4 months
  Measured with Likert scale

SECONDARY OUTCOMES:
Gender differences | 4 months
  to assess gender differences in the use of eHealth

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Ortiz, PhD, MD, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: Undecided
In the near future, we plan to extend the use of the digital care path nationwide. This might allow the participation of other centers in the future.

REFERENCES:
- [Derived] Ortiz F, Grasberger J, Ekstrand A, Helantera I, Giunti G. Interactive Health Technology Tool for Kidney Living Donor Assessment to Standardize the Informed Consent Process: Usability and Qualitative Content Analysis. JMIR Form Res. 2024 Jul 9;8:e47785. doi: 10.2196/47785. PMID 38981119
- [Derived] Ortiz F, Giunti G. Usability assessment of an interactive health technology for kidney living donors: protocol for a prospective cross-sectional survey. BMJ Open. 2022 Jan 3;12(1):e051166. doi: 10.1136/bmjopen-2021-051166. PMID 34980611